CLINICAL TRIAL: NCT04880824
Title: Analysis of the Pathophysiology of Frailty Syndrome and Clinical Development of Frailty Within the Framework of the Innovation Fund Project PRÄP-GO (ANA-PRÄP-GO)
Brief Title: Analysis of Frailty Syndrome Within the Framework of the Innovation Fund Project PRÄP-GO (ANA-PRÄP-GO)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: ANA-PRAEP-GO
Record Dates: First submitted 2021-04-23; First posted 2021-05-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetical analyses from blood samples: Multiplex gene expression analyzes (neuroinflammation and micro RNA panels) and APOE polymorphisms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PG cohort: 800 randomized surgical study patients with a frailty syndrome (Pre-frail and frail) of the intervention study PRÄP-GO (PG cohort). 400 study patients receive the intervention and 400 study patients receive standard of care.
  Interventions: Behavioral: Prehabilitation- new form of care
- NFC cohort: 400 non-frail surgical control group (NFC cohort)
- NO cohort: 300 non-operative control group (NO cohort)
- GB cohort: Skill-Change-Management: a maximum of 30 coworkers and analysis of guiding principle: to a maximum of 35 patients, 30 relatives and 45 coworkers

INTERVENTIONS:
Behavioral: Prehabilitation- new form of care — The participants in the intervention group take part in a shared decision-making (SDM) conference to plan the intervention. The therapeutic content of the prehabilitation is defined individually for each patient in the SDM conference. Prehabilitation will be a structured and individually tailored 3-week program.
  Groups: PG cohort

SUMMARY:
The patients included in PRÄP-GO and the corresponding comparison cohorts will be offered to participate in this complementary study in order to be able to carry out a detailed characterization and phenotyping of the frailty complex.

Amendment vote of 08/05/2024: Recruitment extension of Non-frail surgical control group (NFC cohort) until August 31, 2025.

DETAILED DESCRIPTION:
As part of the innovation fund project PRÄP-GO (EA1/225/19), a multimodal intervention is being conducted in patients with a frailty syndrome. However, the health care research project is limited to evaluating clinical issues only. In order to be able to research further pathophysiological, clinical, psychosocial and work-organizational connections, different groups of participants will be offered the participation in this scientific support program of PRÄP-GO.

The groups of participants in this accompanying program ANA-PRÄP-GO are:

* Randomized study patients with a frailty syndrome of the intervention study PRÄP-GO (PG cohort)
* Non-frail surgical control group (NFC cohort)
* Non-surgical comparison group (NO cohort)
* Participants with health professions (GB cohort)

Additionally, relatives of the patients can be included.

Subprojects are included to reflect research questions of interest in sub groups:

* Success of endoprosthetic implants (clinical outcome and gait pattern after total hip arthroplasty and total knee arthroplasty in frail patients)
* Functional treatment outcome and health-related quality of life after elective spinal surgery in the PG cohort, in the NFC cohort, and in the NO cohort
* Hemodynamic evaluation in patients of the PG and NFC cohort with preoperative abnormal cardiovascular function
* Establishment of a German standard database for 14 CANTAB tests by CANTAB Connect technology
* Aggregated evaluation of the cognitive data of different surgical cohorts from studies carried out at the department of anesthesiology to describe domain-specific changes in the perioperative course
* Perspectives of different health professional groups regarding barriers and facilitators in the implementation of a prehabilitation program and necessary changes in skill, organizational and management, and communication in an interdisciplinary setting
* Perspectives of patients and significant others regarding the organizational pathway of the prehabilitation program
* Frequency, pathophysiology and trajectory of muscle weakness as well as functional impairments of patients admitted to intensive care units of the PG and NFC cohort and their long-term outcomes.
* The gut microbiome as a potential risk factor for perioperative neurocognitive disorders (PNDs) in the elderly
* Evaluation of nutrition data in all cohorts (e.g. adherence to mediterranean diet, nutrition habits, nutritional status, dental status etc.)

ELIGIBILITY:
PG cohort:

Inclusion criteria

* Consent given and inclusion in PRÄP-GO
* Patient capable of giving consent or existing legal guardian in the case of patients not capable of giving consent

Exclusion criteria

- None

NFC cohort:

Inclusion criteria

* Patient capable of giving consent or existing legal guardian in the case of patients not capable of giving consent
* Age ≥ 70 years
* Elective surgery planned
* Expected anesthesia duration> 60 min
* No frailty syndrome (0 positive out of 5 standardized parameters) according to the physical frailty phenotype (Fried et al., 2001)

Exclusion criteria

* Severe cardiac or pulmonary disease (NYHA IV, Gold IV)
* Intracranial interventions
* Moribund patients (palliative situation)
* Patients with a neuropsychiatric clinical picture or severe hearing and / or visual acuity impairment (not compensated by visual or hearing aids), which limit the performance of the neurocognitive tests
* Insufficient language skills
* Participation in another interventional rehabilitation study or a study according to the German Drug Law or the medical Device Law that has not been approved by the study leader (Exception: parallel participation in adjuvant therapy study).

NO cohort:

Inclusion criteria

- Age ≥ 70 years

* No elective surgery planned
* No surgery within 6 months prior to study enrollment

Exclusion criteria - See NFC cohort

GB cohort:

Inclusion criterion

- Doctor, nurse or therapist from the cooperation partners of PRAEP-GO who were involved in the project

Exclusion criterion

- Language barrier

Relatives:

Inclusion criteria

* Member of a patient in the PRÄP-GO cohort
* Age ≥ 18 years

Exclusion criterion

- Language barrier

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The groups of participants in this scientific accompanying program ANA-PRÄP-GO are:
  * Randomized study patients with a frailty syndrome of the intervention study PRÄP-GO (PG cohort)
  * Non-frail surgical control group (NFC cohort)
  * Non-surgical comparison group (NO cohort)
  * Participants with health professions (GB cohort)
  * Relatives of the included patients
Sampling Method: Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Frailty | Up to 1 year
  Frequency of frailty is measured by modified Fried criteria (category 1 +2 = pre-frail, category 3 -5 = frail)
Neuro-cognitive disorder (NCD) | Up to 1 year
  Frequency of neuro-cognitive disorder (mild / major NCD)

SECONDARY OUTCOMES:
Incidence of delirium | During the hospital stay, an expected average of 1 week
  Incidence of delirium, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V), Richmond Agitation Scale (RASS), Nursing Delirium Screening Scale (Nu-DESC), Confusion Assessment Method (CAM), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), along with the delirium severity scores Confusion Assessment Method Severity-Score (CAM-S) in English, Intensive Care Delirium Screening Checklist (ICDSC), Delirium Rating Scale Revised 98 (DRS-R-98) in English and patient chart review. The assessment period is from the recovery room up to five postoperative days or until hospital discharge.
Severity of delirium | During the hospital stay, an expected average of 1 week
  Severity of delirium defined as a composite score based on: Confusion Assessment Method Severity-Score(CAM-S); Confusion Assessment Method (CAM), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Delirium Rating Scale Revised (DSR-R-98) in English, Intensive Care Delirium Screening Checklist (ICDSC) and Nursing Delirium Screening Scale (Nu-DESC) and patient chart review.
Nursing Delirium Screening Scale (Nu-DESC) | During the hospital stay, an expected average of 1 week
  Nursing Delirium Screening Scale (Nu-DESC) score of ≥ 2 is indicative of delirium, range: 0-10 points, 10 = most severe.
Confusion Assessment Method (CAM) | During the hospital stay, an expected average of 1 week
  Confusion Assessment Method (CAM) score is indicative of delirium, if the items 1 and 2 and 3 or the items 1 and 2 and 4 are measured positively.
Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | During the hospital stay, an expected average of 1 week
  Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score is indicative of delirium, if the items 1 and 2 and 3 or the items 1 and 2 and 4 are measured positively.
Confusion Assessment Method Severity-Score (CAM-S Long Form) in English | During the hospital stay, an expected average of 1 week
  The Confusion Assessment Method Severity-Score (CAM-S Long Form) is an 10-item delirium screening instrument (range: 0-19 points, 19 = most severe).
Intensive Care Delirium Screening Checklist (ICDSC) | During the hospital stay, an expected average of 1 week
  The ICDSC is an 8-item delirium screening instrument (range: 0-8 points). The score is indicative of delirium, if the item is > 3.
Delirium Rating Scale Revised 98 in English (DRS-R-98) | During the hospital stay, an expected average of 1 week
  The delirium rating scale revised 98 is a delirium screening instrument (range 0-46). The score is indicative of delirium, if the item is > 14.5.
Delirium Severity Scale (CAM-ICU-7) in English | During the hospital stay, an expected average of 1 week
  A 7-point rating scale (0-7) was derived from the CAM-ICU and RASS assessments 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Number of Participants with Delirium as Determined by Chart Review | During the hospital stay, an expected average of 1 week
  Delirium is identified chart-based.
Delirium days | During the hospital stay, an expected average of 1 week
  The duration of delirium is measured in days.
COVID-19 | Up to 1 year
  SARS-CoV-2 infection
Cardiovascular function 1 | Up to 1 year
  Cardiovascular function is measured by Transesophageal Echocardiography.
Cardiovascular function 2 | Up to 1 year
  Cardiovascular function is measured by cardiovascular complications.
Ethical aspects | Up to 1 year
  Wishes of the patient about the intensity of therapy and therapy goals are measured with a questionnaire.
Patient satisfaction | Up to 1 year
  Patient satisfaction score is measured with a likert scale (0 - 10)
Patient-related outcome measures (PROMS) | Up to 1 year
  Different tools and questionnaires are combined to measure Patient-related outcome.
Patient-related experience measures (PREMS) | Up to 1 year
  Patient-reported experiences of health care are measured with a questionnaire.
Incidence of dementia | Up to 1 year
  incidence of dementia is measured by MOCA
Incidence of cognitive impairment | Up to 1 year
  incidence of cognitive impairment is measured by a validated score.
Findings of Memory consultation | Up to 1 year
  During memory consultation cognitive diagnostic findings are measured.
Stress | Up to 1 year
  Stress is measured by Perceived Stress Questionnaire (PSQ20), which ranges from 20-80 points
Anxiety 1 | Up to 1 year
  Anxiety is measured by Generalized Anxiety Disorder 7, points range from 0-21
Anxiety 2 | Up to 1 year
  Anxiety 2 is measured by Faces Anxiety Scale, a valid single-item for self-report measure of state
Insomnia | Up to 1 year
  Insomnia is measured by Insomnia Severity Index (ISI), which ranges from 0- 21 points
Neuroimaging | Up to 1 year
  Routine neuroimaging results were planned to be documented in the hospital including all techniques to image the nervous system as ultrasound, magnetic resonance imaging, conventional radiography, computed tomography and positron emission tomography.
Demand of health services | Up to 1 year
  The need of treatment for curing an illness.
Adverse events | Up to 1 year
  Adverse events are measured in all participants, who receive study measurements
Nutritional Status | Up to 1 year
  Changes in the nutritional status after elective surgery
Adherence to Mediterranean diet (MD) | Up to 1 year
  Adherence to Mediterranean diet (MD) is measured with a German Medi-Score, could range from 0 to 9, with higher scores (6-9) indicating greater MD adherence.
Sarcopenia | Up to 1 year
  The composite outcome measure "Sarcopenia" is defined by the following three criteria: 1) low muscle strength (hand grip strength), 2) low muscle quantity (calf circumference and 3) low physical performance (gait speed). Criterion (1) identifies probable sarcopenia, additional documentation of criterion (2) confirms sarcopenia diagnosis, and if all criteria (1), (2) and (3) are met, sarcopenia is considered severe.
Calf circumference | Up to 1 year
  Calf circumference is measured in a standardized position and documented in centimeter.
Arm circumference | Up to 1 year
  Arm circumference is measured in a standardized position and documented in centimeter.
Dental status | Up to 1 year
  (number of teeth, Oral Health Assessment Tool (OHAT), Geriatric Oral Health Assessment Index (GO-HAI), questions regarding prothesis, dentist visits and dental care)
Quality of life | Up to 1 year
  Quality of life is measured by Care Related Quality of Life (CarerQoL)
Postoperative complications | Up to 30 days
  Complications are measured according to the Clavien-Dindo classification
Psychometric properties of the Meta Memory questionnaire | During the hospital stay, at the beginning of the investigation, an average of two hours.
  Psychometric properties of the Meta Memory questionnaire are measured twice before surgery.
Number of participants with changes in laboratory values 1 | Up to 1 year
  Routine laboratory results were planned to be documented in the hospital including hemoglobin, lymphocytes, total neutrophils, platelet count and white blood cell (WBC) count from blood samples.
Number of participants with changes in laboratory values 2 | Up to 1 year
  Routine laboratory results were planned to be documented from the general practitioner including hemoglobin, lymphocytes, total neutrophils, platelet count and white blood cell (WBC) count from blood samples.
APOE polymorphisms | Up to 1 year
  APOE polymorphisms are measured from whole blood once during hospital stay, an expected average of one week.
Total interleukin-8 | Up to 1 year
  Total interleukin-8 is measured from whole blood
Cholinesterases 1 | Up to 1 year
  Acetylcholinesterase and Butyrylcholinesterase are measured from liquor
Cholinesterases 2 | Up to 1 year
  Acetylcholinesterase and Butyrylcholinesterase are measured from whole blood
Intracellular pH | Up to 1 year
  Intracellular pH is measured from whole blood.
Autophagy of platelets | Up to 1 year
  Autophagy of platelets is measured from whole blood.
Peripheral Blood Mononuclear Cell | Up to 1 year
  Peripheral Blood Mononuclear Cell are measured from whole blood.
Multiplex gene expression analyzes (neuroinflammation and micro RNA panels) | Up to 1 year
  Multiplex gene expression analyzes (neuroinflammation and micro RNA panels) are measured from whole blood
Autoantibodies | Up to 1 year
  Autoantibodies against beta2-adrenergic receptor, muscarinic acetylcholine receptor (M3 / M4), serotonin receptor, dopamine receptor are measured from serum
Trypotophan metabolites and short-chain fatty acids | Up to 1 year
  Trypotophan metabolites and short-chain fatty acids are measured from serum with metabolomic analysis
Biomarker panel | Up to 1 year
  Biomarker are measured from serum by metabolomic analyses to characterize the frailty complex.
Cytokines | Up to 1 year
  Cytokines (IFN-Ɣ IL-1β IL-4 IL-6 IL-10 IL-17A IL-17E IL-17F IL-21 IL-23 TGF-β1) are measured from plasma
Chemokines | Up to 1 year
  Chemokines (CCL2 (MCP-1) CCL3 CCL4 CCL5 (RAN-TES) CCL11 (Eotaxin) CCL19 CCL20 CXCL1 CXCL8 (IL-8) CXCL10 (IP-10) CXCL12 (SDF1A) are measured from plasma
Markers immune-brain axis and gut-brain axis | Up to 1 year
  Markers immune-brain axis and gut-brain axis (zonulin, endothelial cell-specific molecule 1, S100A6, S100A8, S100A9, S100P, S100beta, Interleu-kin-16, CD162, BDNF, CD272, p-selectin, be-ta2microglobulin , Haptoglobin, cathelicidin, NCAM-1, BTLA and CXCR5) are measured from plasma
Protein panel | Up to 1 year
  Proteins are measured from plasma by proteome analysis.
Microbiome 1 | Up to 1 year
  Analyzes of bacteria-specific 16S DNA from different biomaterial.
Microbiome 2 | Up to 1 year
  Analyzes of sequences of known microorganisms from different biomaterial.
Serum albumin | Up to 1 year
  Serum albumin is measured from whole blood
HbA1c | Up to 1 year
  HbA1c is measured from whole blood
Vitamin D (cholecalciferol) | Up to 1 year
  Vitamin D is measured from whole blood
Dementia markers | Up to 1 year
  Dementia markers: beta amyloid 1-40, beta-amyloid 1-42, beta-amyloid ratio (42/40 * 10), phospho-TAU, protein 14-3-3, PRPSc, TAU (total tau) are measured from liquor
Analysis of microbiome | Up to 1 year
  Microbial diversity is measured from blood, urine and feces (e.g. Shannon index)
Analysis of urine | Up to 1 year
  Relative frequency of metabolites is measured in urine
Biobanks samples | Up to 1 year
  Secondary use of the biological samples in particular for research purposes
Hip Osteoarthritis Outcome | Up to 1 year
  Hip Osteoarthritis Outcome is measured from Hip disability and Osteoarthritis Outcome Score (HOOS) in orthopedic patients from PG cohort
Knee Osteoarthritis Outcome | Up to 1 year
  Knee Osteoarthritis Outcome is measured from Knee injury and Osteoarthritis Outcome (KOOS) in orthopedic patients from PG cohort
Gait analysis 1 | Up to 1 year
  Temporal (e.g.: total activity duration, stance time) parameters are measured in orthopedic patients from PG cohort.
Gait analysis 2 | Up to 1 year
  Kinetic parameters (e.g.: vertical plantar loading, loading symmetry) are measured in orthopedic patients from PG cohort.
Range of Motion of the hip/knee | Up to 1 year
  Range of Motion of the hip/knee is measured during orthopedic investigation of PG cohort patients
Hip abduction force (for total hip arthroplasty patients) | Up to 1 year
  Hip abduction force is measured during orthopedic investigation of PG cohort patients
Knee extension and flexion force measurement (for total knee arthroplasty patients) | Up to 1 year
  Knee extension and flexion force measurement is measured during orthopedic investigation of PG cohort patients
Clinical investigation | Up to 1 year
  Clinical investigation is measured by a neurosurgical method in patients from PG and NFC cohorts who undergo elective spine surgery and in control patients from NO cohort
Oswestry disability index (ODI) | Up to 1 year
  ODI is measured in patients from PG and NFC cohorts who undergo elective spine surgery and in control patients from NO cohort.
Back pain | Up to 1 year
  Low Back pain is measured by the Roland Morris Low Back pain and disability questionnaire in patients (PG, NFC, NO cohorts) with lumbal spine problems.
Leg pain | Up to 1 year
  Leg pain is measured by 100mm visual analog scale in patients (PG, NFC, NO cohorts) with lumbal spine problems.
Sciatica Bothersomeness Index | Up to 1 year
  To establish values for paresthesia, weakness and leg pain the Sciatica Bothersomeness Index is measured n patients (PG, NFC, NO cohorts) with lumbal spine problems.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | Up to 1 year
  To measure Disabilities of the Arm, Shoulder and Hand the DASH questionnaire is used in patient (PG, NFC, NO cohort) in patients with cervical spine problems
Modified Japanese orthopaedic association scale | Up to 1 year
  The modified Japanese Orthopaedic Association scale is used to establish criteria for mild, moderate and severe impairment in patients with degenerative cervical myelopathy in patients (PG, NFC, NO cohorts) with cervical spine problems
ASIA Impairment Scale (AIS) | Up to 1 year
  ASIA Impairment Scale is used to measure for patients with spinal myelopathies or spinal cord injuries in patients from PG and NFC cohorts who undergo elective spine surgery and in control patients from NO cohort
Skill management | Up to 1 year
  Multiprofessional skill management is evaluated in all participating occupations of the GB cohort in qualitative interviews.
Acceptance of participatory decision-making | Up to 1 year
  Acceptance of participatory decision-making before and after participating in an SDM conference.
Depth of anesthesia | During surgery, an expected average of 2 hours
  Depth of anesthesia is measured by brainwaves in different patient states which range from awake, sedated, unresponsive, surgically anesthetized to deeply anesthetized.
Electroencephalography spectral analysis | During the hospital stay, at the beginning of the investigation, an average of one hour.
  Electroencephalography spectral analysis is measured by brainwaves preoperatively.
Electroencephalography band power | During the hospital stay, an expected average of 1 week
  Electroencephalography band power is measured postoperatively by an electroencephalography monitor at postoperative day 3 in all patients and in patients with delirium until 48 hours without positive delirium screening
Effect of analgesics | During the hospital stay, an expected average of 1 week
  Pain is evaluated with the Dolosys Paintracker. The Paintracker is a handy monitoring device to determine the analgesia needed for patients based on the pain reflex technique.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (27):
- Germany (27):
  - Praxis Prof. Dr med. Ulrich Schwantes, Schwante, Brandenburg
  - Charité-Universitätsmedizin Berlin, Department of Physical Medicine, Berlin
  - Praxis Landgraf, Berlin
  - Department of Anesthesiology and Operative Intensive Care Medicine (CBF), Berlin
  - Department of Anesthesiology and Intensive Care Medicine, Charité - University Medicine, Berlin
  - Paul Gerhard Diakonie - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Paul Gerhard Diakonie - Evangelisches Krankenhaus Hubertus, Berlin
  - Paul Gerhard Diakonie - Martin-Luther-Krankenhaus, Berlin
  - Auguste-Viktoria-Klinikum - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - CARITAS Klinik Maria Heimsuchung, Berlin
  - Dominikus-Krankenhaus, Berlin
  - Humboldt-Klinikum - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Klinikum im Friedrichshain - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Sankt Jospeph Krankenhaus, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Universitätsklinikum Mannheim GmbH, Berlin
  - Wenckebach-Klinikum - Vivantes - Netzwerk für Gesundheit GmbH, Berlin
  - Carl-Thiem-Klinikum, Cottbus
  - Werner Forßmann-Krankenhaus, Eberswalde
  - Klinikum Frankfurt Oder GmbH, Frankfurt (Oder)
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinikum Harburg, Harburg
  - Sana Kliniken Sommerfeld, Kremmen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Universität zu Lübeck, Lübeck
  - Klinikum der Universität München, LMU Campus Großhadern, München
  - Klinikum rechts der Isar - Technische Universität München, München
  - München Klinik Bogenhausen, München

IPD SHARING:
Plan to Share IPD: No